CLINICAL TRIAL: NCT07355712
Title: Combined Effect of Prolotherapy and Personalized Physical Activity on Knee Osteoarthritis Progression, Impact on IL-1β, MMP-3 Biomarkers and Clinical Outcomes
Brief Title: Combined Effect of Prolotherapy and Personalized Physical Activity on Knee Osteoarthritis Progression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: Faculty of Medicine, Gadjah Mada University (Unknown); Universitas Islam Indonesia (Other)
Responsible Party: Principal Investigator, muhammad yusuf hisam, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KE/FK/1000/EC/2024; s3 fkkmk ugm (Other: FKKMK UGM)
Record Dates: First submitted 2025-11-25; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Prolotherapy
Keywords: Knee Osteoarthritides; Prolotherapy; physical activity; interleukin-1beta; matrix Metalloproteinase 3
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Prolotherapy

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention (prolotherapy combined with physical activity or prolotherapy alone) within the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolotherapy + Personalized Physical Activity Program (Experimental): This arm will be using prolotherapy with 20 mL of 15% hypertonic dextrose solutions and 2 mL of 2% lidocaine and physical therapy starting 2 day post-injection with guidance of trained professionals and exercise educational videos supplementation (10 repetitions per session, 3 sessions per day, 3 days per week)
  Interventions: Combination Product: Prolotherapy; Other: Personalized Physical Activity Program
- Prolotherapy Only (Active Comparator): This arm will be using prolotherapy with 20 mL of 15% hypertonic dextrose solutions and 2 mL of 2% lidocaine
  Interventions: Procedure: Prolotherapy Only

INTERVENTIONS:
Procedure: Prolotherapy Only — This arm will be using prolotherapy with 20 mL of 15% hypertonic dextrose solutions and 2 mL of 2% lidocaine
  Arms: Prolotherapy Only
Combination Product: Prolotherapy — This arm will be using prolotherapy with 20 mL of 15% hypertonic dextrose solutions and 2 mL of 2% lidocaine
  Arms: Prolotherapy + Personalized Physical Activity Program
Other: Personalized Physical Activity Program — A physical therapy program starting 2 day post-injection with guidance of trained professionals and exercise educational videos supplementation (10 repetitions per session, 3 sessions per day, 3 days per week)
  Arms: Prolotherapy + Personalized Physical Activity Program

SUMMARY:
The aim of this clinical trial is to assess whether prolotherapy combined with personal physical activity is effective in managing pain (measured using the VAS and WOMAC scales) and improving the quality of life in participants with Grade 2 Knee Osteoarthritis (OA).

This trial will also measure the levels of IL-1β and MMP-3 in the participants. The primary research questions are:

1. Does prolotherapy combined with personal physical activity reduce pain levels and improve clinical outcomes in participants with knee OA compared to those receiving prolotherapy ?
2. How does this intervention affect the levels of IL-1β and MMP-3 in participants?

Researchers will compare prolotherapy combined with personal physical activity to prolotherapy alone to determine its impact on clinical outcomes and changes in biomarkers in patients with knee OA.

DETAILED DESCRIPTION:
The objective of this clinical trial is to evaluate the levels of IL-1β and MMP-3, clinical outcomes related to pain (measured using the Visual Analog Scale (VAS) and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)), as well as the quality of life in participants with knee osteoarthritis (OA) who are treated with pain management through prolotherapy combined with personalized physical activity. This trial aims to develop a complementary therapy or an alternative treatment option that is cost-effective, accessible, and potentially more affordable for the broader population.

Study Design/Methods:

This study will utilize a Randomized Controlled Trial (RCT) design with pre- and post-test assessments.

Group/Arm :

* Experimental Group (Prolotherapy and Personalized Physical Activity Program)
* Active Comparator/Control (Prolotherapy only)

Intervention :

* Experimental Group: using prolotherapy with 20 mL of 15% hypertonic dextrose solutions and 2 mL of 2% lidocaine and physical therapy starting 2 days post-injection with guidance of trained professionals and exercise educational videos (10 repetitions per session, 3 sessions per day, 3 days per week)
* Active Comparator Group: using prolotherapy with 20 mL of 15% hypertonic dextrose solutions and 2 mL of 2% lidocaine

Measurement :

* The primary outcome will be a clinical assessment measured using theWOMAC questionnaire and VAS
* The secondary outcome will be biomarker data of IL-1 Beta and MMP-3 measured with ELISA using kits from ABclonal, IL-1Beta (Cat. No. RK00001, Lot No. 9680034260724) and MMP-3 (Cat. No. RK00308, Lot No. 9680000230724).

Data Analysis Plan:

The data will be analyzed using the Kappa Test, Univariate Analysis, and Bivariate Analysis (Independent T-Test, Paired T-Test, Wilcoxon Test, Chi-Square, Spearman and Pearson Correlation Tests, and ANCOVA).

Anticipated Outcomes:

* Low risk of allergies
* Reduction in pain levels in participants
* Improvement in functional outcomes of participants

Risk and Benefit:

Risks:

- Possible side effects or complications, such as allergic reactions or infections, may occur during the study.

Benefits:

- This study seeks to identify a new and effective alternative therapy and complementary treatment that is more affordable and widely accessible. It is expected to provide significant pain relief, functional improvements, and enhanced quality of life for patients suffering from knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with primary knee osteoarthritis (OA) diagnosed by ultrasonography who provided written informed consent.
* Participants were required to be cooperative and capable of complying with the study protocol

Exclusion Criteria:

* A history of traumatic knee arthritis
* Knee OA associated with trauma, fracture, ankylosing spondylitis, or septic arthritis
* Major comorbidities significantly impairing quality of life (e.g., cancer, heart failure, renal failure, stroke)
* Use of NSAIDs or systemic steroids within 1 week
* Intra-articular corticosteroid injection within 2 months; or current use of injectable or hormonal contraception.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Pain and Functional Capacity | 6 week
  The primary outcome measure for this study is pain dan functional capacity using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
  WOMAC Questionnaire consist of 3 subscales (pain, stiffness, and physical function). Pain subscale can be scored between 0-20 points, stiffness subscale can be scored between 0-8 points, and physical function subscales can be scored between 0-68 points. Those points can be interpreted better if its low and worser if it high in total (0-24 points for mild, 25-48 points for moderate, and 49-72 points for severe)

SECONDARY OUTCOMES:
Concentration of IL-1 Beta and MMP-3 | 6 week
  Biomarker such IL-1 Beta and MMP-3 were measured by ELISA using kits from ABclonal (Cat. No. RK00001, Lot No. 9680034260724 for IL-1 Beta) and (Cat. No. RK00001, Lot No. 9680034260724 for MMP-3)
Pain with Visual Analog Scale | 6 weeks
  VAS Questionnaire points will be between 0 (no pain) and 100 (severe intolerable pain)
Quality of Life with EQ-5D-5L | 6 weeks
  EQ-5D-5L Indonesian value set will have 5 segments (mobility, looking after myself, doing usual activities, pain and discomfort, feeling worried, sad, or unhappy), each segments will have 0-5 points The points can be interpret as if the higher the points, the better quality of life will be

CONTACTS AND LOCATIONS:
Overall Officials: muhammad yusuf hisam MYH Hisam, MD, Principal Investigator — Gadjah Mada University
Locations (1):
- fkkmk UGM, Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT07355712/Prot_000.pdf
  • Informed Consent Form (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT07355712/ICF_001.pdf